CLINICAL TRIAL: NCT04512911
Title: Endocardial-Epicardial Radiofrequency Ablation of Ventricular Tachycardia in Patients With Ischemic Cardiomyopathy
Brief Title: Comparison of Ventricular Tachycardia Ablation Strategies in Patients With Ischemic Cardiomyopathy
Acronym: EPI-VT
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: IRB approval expired 1/23/2023 and eclipsed the 6 month institutional window where study can be reinitiated via progress report. No enrollment has taken place.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-10639
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Ventricular Tachycardia
Keywords: Ventricular tachycardia; Catheter ablation; Epicardial ablation; arrhythmia recurrence
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: A total of 100 patients will be randomized in 1:1 fashion to investigation arms Endocardial - Epicardial (20 patients) or Endocardial ablation (20 patients) if patients have previously failed AAD and in 1:1:1 fashion randomization to Endocardial - Epicardial ablation (20 patients), Endocardial ablation (20 patients) and AAD (20 patients) if patients have not failed AAD previously. If during follow up VT recurrence occurs, treatment method that patient was assigned to will be considered failed and patients will undergo redo ablation (same as previously assigned to) or if AAD failed patient will be added a second AAD or changed to another AAD. If during follow up after second procedure or adjustment of AAD patient experiences VT recurrence the treatment method will be considered failed.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the ablation procedures and medications treatment assignment, physicians and patients cannot be blinded to the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patients who didn't fail AAD (Active Comparator): This group of patients will be randomized to 3 subgroups: 1) Endocardial ablation; 2) Endocardial - Epicardial ablation; 3) Antiarrhythmic medications
  Interventions: Procedure: Endocardial ablation; Procedure: Endocardial- Epicardial ablation; Drug: Antiarrhythmic medications
- Patients who failed AAD (Active Comparator): This group of patients will be randomized to 2 subgroups: 1) Endocardial ablation; 2) Endocardial - Epicardial ablation
  Interventions: Procedure: Endocardial ablation; Procedure: Endocardial- Epicardial ablation

INTERVENTIONS:
Procedure: Endocardial ablation — Endocardial ablation of VT
Procedure: Endocardial- Epicardial ablation — Epicardial ablation of VT in addition to endocardial ablation
Drug: Antiarrhythmic medications — Addition of anti arrhythmic medication or dose increase
  Arms: Patients who didn't fail AAD

SUMMARY:
This is a prospective multicenter randomized open-label study aiming to assess whether endocardial or endocardial-epicardial ablation is superior to the standard approach (i.e., Antiarrhythmic drugs) in achievement of long-term ventricular tachycardia (VT) treatment success.

DETAILED DESCRIPTION:
Comparison of Ventricular Tachycardia Ablation Strategies in Patients With Ischemic Cardiomyopathy (EPI VT) is a prospective multicenter randomized controlled study that is planned as a pilot study to include 100 patients. The aim of our study is to assess whether endocardial or endocardial-epicardial ablation is superior to the standard approach (i.e., Antiarrhythmic drugs) in the achievement of long-term ventricular tachycardia (VT) treatment success. Patients will be stratified into two groups depending on the history of taking antiarrhythmic medications (AAD) and each group will be further randomized 1:1 for endocardial and epicardial ablation vs endocardial only ablation in group who failed AAD. And in the group who didn't fail AADs patients will be randomized 1:1:1 into 3 groups: endocardial and epicardial ablation, endocardial only ablation or antiarrhythmic medications. Follow up planned at 3, 6 and 12 months, if VT recurrence is noted, repeated procedure (according to initially allocated group) or adjustment of medications (if AAD group) will be performed. Follow up at 3, 6 and 12 months is also planned after a repeat procedure/ medications adjustment.

Primary endpoints include freedom from documented VT episodes (> 30 seconds) at 12 months after the first ablation procedure or on antiarrhythmic medication and freedom from documented VT episodes (>30 seconds) at 12 months after the second ablation procedure or on two antiarrhythmics combined.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 or greater
* Patient with ≥ 1 episode of VT (i.e., Sustained VT more than 30 seconds or VT with any ICD therapy)
* Patients with ischemic cardiomyopathy, EF less than 50%, documented history of CAD

Exclusion Criteria:

* Patients with ventricular fibrillation.
* Reversible causes of VT.
* Patients with contraindications to systemic anticoagulation with heparin or coumadin, direct thrombin inhibitor or factor Xa inhibitors.
* Patients with prior procedure involving opening the pericardium or entering the pericardial space (e.g., CABG, heart transplantation, valve surgery) were adhesions are suspected
* Any prior ablation for the ventricles or any prior epicardial ablation
* Documented history of myocardial infarction within 1 month prior to the planned study intervention
* Documented symptomatic carotid disease defined as > 70% stenosis or > 50% stenosis with symptoms
* Any history of thoracic radiation with the exception of localized radiation treatment for breast cancer
* Active pericarditis
* Active endocarditis\Any documented history or autoimmune disease associated with pericarditis
* Thrombocytopenia (platelet count < 100 x 109/L)
* Body Mass Index (BMI > 45)
* Patients who are pregnant.

  1. Pregnancy will be assessed by urine pregnancy testing prior to the ablation procedure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-01-23 (Estimated); Study Completion 2023-01-23 (Estimated)

PRIMARY OUTCOMES:
Freedom from documented VT episodes | 12 months
  Freedom from documented VT episodes (greater than 30 seconds) at 12 months after the first ablation procedure or on antiarrhythmic medication.
Freedom from documented VT episodes after second intervention | 12 months after second intervention
  Freedom from documented VT episodes (greater than 30 seconds) at 12 months after the second ablation procedure or on two antiarrhythmics combined.

SECONDARY OUTCOMES:
Incidence of peri-procedural and 12-month post procedural complications, | 12 months
  These complications include but not limited to ischemic stroke, cardiac perforation, rehospitalization, and death.
Procedure duration and fluoroscopy time | Up to 4 hours (During ablation procedure)
  Procedure duration and fluoroscopy time
Number of repeat procedures | 12, 24 months
  Number of repeat ablations
Cost-effectiveness analysis | 12 months
  The CEA will examine the cost of health care resources and health outcomes from the ablation procedure to 1-year postoperatively. The costs will include all health care utilization during this time. Health care utilization, and associated costs, related to the patients' condition, the procedure and adverse events will be the basis of a sensitivity analysis.
Long-term follow-up to evaluate freedom of documented VT episodes | 24 and 60 months
  Long-term follow-up at 24 and 60 months to evaluate freedom of documented VT episodes (>30 seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Romero, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine; Luigi Di Biase, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, Cardiology, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Connolly SJ, Hallstrom AP, Cappato R, Schron EB, Kuck KH, Zipes DP, Greene HL, Boczor S, Domanski M, Follmann D, Gent M, Roberts RS. Meta-analysis of the implantable cardioverter defibrillator secondary prevention trials. AVID, CASH and CIDS studies. Antiarrhythmics vs Implantable Defibrillator study. Cardiac Arrest Study Hamburg . Canadian Implantable Defibrillator Study. Eur Heart J. 2000 Dec;21(24):2071-8. doi: 10.1053/euhj.2000.2476. PMID 11102258
- [Background] Poole JE, Johnson GW, Hellkamp AS, Anderson J, Callans DJ, Raitt MH, Reddy RK, Marchlinski FE, Yee R, Guarnieri T, Talajic M, Wilber DJ, Fishbein DP, Packer DL, Mark DB, Lee KL, Bardy GH. Prognostic importance of defibrillator shocks in patients with heart failure. N Engl J Med. 2008 Sep 4;359(10):1009-17. doi: 10.1056/NEJMoa071098. PMID 18768944
- [Background] Tung R, Vaseghi M, Frankel DS, Vergara P, Di Biase L, Nagashima K, Yu R, Vangala S, Tseng CH, Choi EK, Khurshid S, Patel M, Mathuria N, Nakahara S, Tzou WS, Sauer WH, Vakil K, Tedrow U, Burkhardt JD, Tholakanahalli VN, Saliaris A, Dickfeld T, Weiss JP, Bunch TJ, Reddy M, Kanmanthareddy A, Callans DJ, Lakkireddy D, Natale A, Marchlinski F, Stevenson WG, Della Bella P, Shivkumar K. Freedom from recurrent ventricular tachycardia after catheter ablation is associated with improved survival in patients with structural heart disease: An International VT Ablation Center Collaborative Group study. Heart Rhythm. 2015 Sep;12(9):1997-2007. doi: 10.1016/j.hrthm.2015.05.036. Epub 2015 May 30. PMID 26031376
- [Background] Bardy GH, Lee KL, Mark DB, Poole JE, Packer DL, Boineau R, Domanski M, Troutman C, Anderson J, Johnson G, McNulty SE, Clapp-Channing N, Davidson-Ray LD, Fraulo ES, Fishbein DP, Luceri RM, Ip JH; Sudden Cardiac Death in Heart Failure Trial (SCD-HeFT) Investigators. Amiodarone or an implantable cardioverter-defibrillator for congestive heart failure. N Engl J Med. 2005 Jan 20;352(3):225-37. doi: 10.1056/NEJMoa043399. PMID 15659722
- [Background] Sapp JL, Wells GA, Parkash R, Stevenson WG, Blier L, Sarrazin JF, Thibault B, Rivard L, Gula L, Leong-Sit P, Essebag V, Nery PB, Tung SK, Raymond JM, Sterns LD, Veenhuyzen GD, Healey JS, Redfearn D, Roux JF, Tang AS. Ventricular Tachycardia Ablation versus Escalation of Antiarrhythmic Drugs. N Engl J Med. 2016 Jul 14;375(2):111-21. doi: 10.1056/NEJMoa1513614. Epub 2016 May 5. PMID 27149033
- [Background] Romero J, Cerrud-Rodriguez RC, Di Biase L, Diaz JC, Alviz I, Grupposo V, Cerna L, Avendano R, Tedrow U, Natale A, Tung R, Kumar S. Combined Endocardial-Epicardial Versus Endocardial Catheter Ablation Alone for Ventricular Tachycardia in Structural Heart Disease: A Systematic Review and Meta-Analysis. JACC Clin Electrophysiol. 2019 Jan;5(1):13-24. doi: 10.1016/j.jacep.2018.08.010. Epub 2018 Sep 26. PMID 30678778
- [Background] Arenal A, Hernandez J, Calvo D, Ceballos C, Atea L, Datino T, Atienza F, Gonzalez-Torrecilla E, Eidelman G, Miracle A, Avila P, Bermejo J, Fernandez-Aviles F. Safety, long-term results, and predictors of recurrence after complete endocardial ventricular tachycardia substrate ablation in patients with previous myocardial infarction. Am J Cardiol. 2013 Feb 15;111(4):499-505. doi: 10.1016/j.amjcard.2012.10.031. Epub 2012 Dec 8. PMID 23228925
- [Background] Tschabrunn CM, Roujol S, Nezafat R, Faulkner-Jones B, Buxton AE, Josephson ME, Anter E. A swine model of infarct-related reentrant ventricular tachycardia: Electroanatomic, magnetic resonance, and histopathological characterization. Heart Rhythm. 2016 Jan;13(1):262-73. doi: 10.1016/j.hrthm.2015.07.030. Epub 2015 Jul 28. PMID 26226214
- [Background] Acosta J, Fernandez-Armenta J, Penela D, Andreu D, Borras R, Vassanelli F, Korshunov V, Perea RJ, de Caralt TM, Ortiz JT, Fita G, Sitges M, Brugada J, Mont L, Berruezo A. Infarct transmurality as a criterion for first-line endo-epicardial substrate-guided ventricular tachycardia ablation in ischemic cardiomyopathy. Heart Rhythm. 2016 Jan;13(1):85-95. doi: 10.1016/j.hrthm.2015.07.010. Epub 2015 Jul 9. PMID 26165946
- [Background] Arenal A, Perez-David E, Avila P, Fernandez-Portales J, Crisostomo V, Baez C, Jimenez-Candil J, Rubio-Guivernau JL, Ledesma-Carbayo MJ, Loughlin G, Bermejo J, Sanchez-Margallo FM, Fernandez-Aviles F. Noninvasive identification of epicardial ventricular tachycardia substrate by magnetic resonance-based signal intensity mapping. Heart Rhythm. 2014 Aug;11(8):1456-64. doi: 10.1016/j.hrthm.2014.04.022. Epub 2014 Apr 16. PMID 24747421
- [Background] Di Biase L, Santangeli P, Burkhardt DJ, Bai R, Mohanty P, Carbucicchio C, Dello Russo A, Casella M, Mohanty S, Pump A, Hongo R, Beheiry S, Pelargonio G, Santarelli P, Zucchetti M, Horton R, Sanchez JE, Elayi CS, Lakkireddy D, Tondo C, Natale A. Endo-epicardial homogenization of the scar versus limited substrate ablation for the treatment of electrical storms in patients with ischemic cardiomyopathy. J Am Coll Cardiol. 2012 Jul 10;60(2):132-41. doi: 10.1016/j.jacc.2012.03.044. PMID 22766340
- [Background] Pokushalov E, Romanov A, Turov A, Artyomenko S, Shirokova N, Karaskov A. Percutaneous epicardial ablation of ventricular tachycardia after failure of endocardial approach in the pediatric population with arrhythmogenic right ventricular dysplasia. Heart Rhythm. 2010 Oct;7(10):1406-10. doi: 10.1016/j.hrthm.2010.06.020. Epub 2010 Jun 17. PMID 20601157
- [Background] Lunati M, Gasparini M, Bocchiardo M, Curnis A, Landolina M, Carboni A, Luzzi G, Zanotto G, Ravazzi P, Magenta G, Denaro A, Distefano P, Grammatico A; InSync ICD Italian Registry Investigators. Clustering of ventricular tachyarrhythmias in heart failure patients implanted with a biventricular cardioverter defibrillator. J Cardiovasc Electrophysiol. 2006 Dec;17(12):1299-306. doi: 10.1111/j.1540-8167.2006.00618.x. PMID 17239095
- [Background] Dorian P, Borggrefe M, Al-Khalidi HR, Hohnloser SH, Brum JM, Tatla DS, Brachmann J, Myerburg RJ, Cannom DS, van der Laan M, Holroyde MJ, Singer I, Pratt CM; SHock Inhibition Evaluation with azimiLiDe (SHIELD) Investigators. Placebo-controlled, randomized clinical trial of azimilide for prevention of ventricular tachyarrhythmias in patients with an implantable cardioverter defibrillator. Circulation. 2004 Dec 14;110(24):3646-54. doi: 10.1161/01.CIR.0000149240.98971.A8. Epub 2004 Nov 8. PMID 15533855
- [Background] Frankel DS, Mountantonakis SE, Robinson MR, Zado ES, Callans DJ, Marchlinski FE. Ventricular tachycardia ablation remains treatment of last resort in structural heart disease: argument for earlier intervention. J Cardiovasc Electrophysiol. 2011 Oct;22(10):1123-8. doi: 10.1111/j.1540-8167.2011.02081.x. Epub 2011 May 3. PMID 21539642
- [Background] Dinov B, Arya A, Bertagnolli L, Schirripa V, Schoene K, Sommer P, Bollmann A, Rolf S, Hindricks G. Early referral for ablation of scar-related ventricular tachycardia is associated with improved acute and long-term outcomes: results from the Heart Center of Leipzig ventricular tachycardia registry. Circ Arrhythm Electrophysiol. 2014 Dec;7(6):1144-51. doi: 10.1161/CIRCEP.114.001953. Epub 2014 Sep 27. PMID 25262159
- [Background] Romero J, Stevenson WG, Fujii A, Kapur S, Baldinger SH, Mehta NK, John RM, Michaud GF, Epstein LM, Koplan BA, Tedrow UB, Kumar S. Impact of Number of Oral Antiarrhythmic Drug Failures Before Referral on Outcomes Following Catheter Ablation of Ventricular Tachycardia. JACC Clin Electrophysiol. 2018 Jun;4(6):810-819. doi: 10.1016/j.jacep.2018.01.016. Epub 2018 Mar 28. PMID 29929675
- [Background] Di Biase L, Burkhardt JD, Pelargonio G, Dello Russo A, Casella M, Santarelli P, Horton R, Sanchez J, Gallinghouse JG, Al-Ahmad A, Wang P, Cummings JE, Schweikert RA, Natale A. Prevention of phrenic nerve injury during epicardial ablation: comparison of methods for separating the phrenic nerve from the epicardial surface. Heart Rhythm. 2009 Jul;6(7):957-61. doi: 10.1016/j.hrthm.2009.03.022. Epub 2009 Mar 19. PMID 19560084
- [Background] Sacher F, Roberts-Thomson K, Maury P, Tedrow U, Nault I, Steven D, Hocini M, Koplan B, Leroux L, Derval N, Seiler J, Wright MJ, Epstein L, Haissaguerre M, Jais P, Stevenson WG. Epicardial ventricular tachycardia ablation a multicenter safety study. J Am Coll Cardiol. 2010 May 25;55(21):2366-72. doi: 10.1016/j.jacc.2009.10.084. PMID 20488308
- [Background] Bai R, Patel D, Di Biase L, Fahmy TS, Kozeluhova M, Prasad S, Schweikert R, Cummings J, Saliba W, Andrews-Williams M, Themistoclakis S, Bonso A, Rossillo A, Raviele A, Schmitt C, Karch M, Uriarte JA, Tchou P, Arruda M, Natale A. Phrenic nerve injury after catheter ablation: should we worry about this complication? J Cardiovasc Electrophysiol. 2006 Sep;17(9):944-8. doi: 10.1111/j.1540-8167.2006.00536.x. Epub 2006 Jun 27. PMID 16800858
- [Background] Cassidy DM, Vassallo JA, Buxton AE, Doherty JU, Marchlinski FE, Josephson ME. The value of catheter mapping during sinus rhythm to localize site of origin of ventricular tachycardia. Circulation. 1984 Jun;69(6):1103-10. doi: 10.1161/01.cir.69.6.1103. PMID 6713614
- [Background] Cassidy DM, Vassallo JA, Miller JM, Poll DS, Buxton AE, Marchlinski FE, Josephson ME. Endocardial catheter mapping in patients in sinus rhythm: relationship to underlying heart disease and ventricular arrhythmias. Circulation. 1986 Apr;73(4):645-52. doi: 10.1161/01.cir.73.4.645. PMID 3948367
- [Background] Kienzle MG, Miller J, Falcone RA, Harken A, Josephson ME. Intraoperative endocardial mapping during sinus rhythm: relationship to site of origin of ventricular tachycardia. Circulation. 1984 Dec;70(6):957-65. doi: 10.1161/01.cir.70.6.957. PMID 6499152
- [Background] Marchlinski FE, Callans DJ, Gottlieb CD, Zado E. Linear ablation lesions for control of unmappable ventricular tachycardia in patients with ischemic and nonischemic cardiomyopathy. Circulation. 2000 Mar 21;101(11):1288-96. doi: 10.1161/01.cir.101.11.1288. PMID 10725289
- [Background] Reddy VY, Neuzil P, Taborsky M, Ruskin JN. Short-term results of substrate mapping and radiofrequency ablation of ischemic ventricular tachycardia using a saline-irrigated catheter. J Am Coll Cardiol. 2003 Jun 18;41(12):2228-36. doi: 10.1016/s0735-1097(03)00492-3. PMID 12821253
- [Background] Arenal A, Glez-Torrecilla E, Ortiz M, Villacastin J, Fdez-Portales J, Sousa E, del Castillo S, Perez de Isla L, Jimenez J, Almendral J. Ablation of electrograms with an isolated, delayed component as treatment of unmappable monomorphic ventricular tachycardias in patients with structural heart disease. J Am Coll Cardiol. 2003 Jan 1;41(1):81-92. doi: 10.1016/s0735-1097(02)02623-2. PMID 12570949
- [Background] Di Biase L, Burkhardt JD, Lakkireddy D, Carbucicchio C, Mohanty S, Mohanty P, Trivedi C, Santangeli P, Bai R, Forleo G, Horton R, Bailey S, Sanchez J, Al-Ahmad A, Hranitzky P, Gallinghouse GJ, Pelargonio G, Hongo RH, Beheiry S, Hao SC, Reddy M, Rossillo A, Themistoclakis S, Dello Russo A, Casella M, Tondo C, Natale A. Ablation of Stable VTs Versus Substrate Ablation in Ischemic Cardiomyopathy: The VISTA Randomized Multicenter Trial. J Am Coll Cardiol. 2015 Dec 29;66(25):2872-2882. doi: 10.1016/j.jacc.2015.10.026. PMID 26718674
- [Background] Jais P, Maury P, Khairy P, Sacher F, Nault I, Komatsu Y, Hocini M, Forclaz A, Jadidi AS, Weerasooryia R, Shah A, Derval N, Cochet H, Knecht S, Miyazaki S, Linton N, Rivard L, Wright M, Wilton SB, Scherr D, Pascale P, Roten L, Pederson M, Bordachar P, Laurent F, Kim SJ, Ritter P, Clementy J, Haissaguerre M. Elimination of local abnormal ventricular activities: a new end point for substrate modification in patients with scar-related ventricular tachycardia. Circulation. 2012 May 8;125(18):2184-96. doi: 10.1161/CIRCULATIONAHA.111.043216. Epub 2012 Apr 4. PMID 22492578
- [Background] Vergara P, Trevisi N, Ricco A, Petracca F, Baratto F, Cireddu M, Bisceglia C, Maccabelli G, Della Bella P. Late potentials abolition as an additional technique for reduction of arrhythmia recurrence in scar related ventricular tachycardia ablation. J Cardiovasc Electrophysiol. 2012 Jun;23(6):621-7. doi: 10.1111/j.1540-8167.2011.02246.x. Epub 2012 Apr 4. PMID 22486970
- [Background] Tung R, Mathuria NS, Nagel R, Mandapati R, Buch EF, Bradfield JS, Vaseghi M, Boyle NG, Shivkumar K. Impact of local ablation on interconnected channels within ventricular scar: mechanistic implications for substrate modification. Circ Arrhythm Electrophysiol. 2013 Dec;6(6):1131-8. doi: 10.1161/CIRCEP.113.000867. Epub 2013 Oct 25. PMID 24162832
- [Background] Briceno DF, Romero J, Villablanca PA, Londono A, Diaz JC, Maraj I, Batul SA, Madan N, Patel J, Jagannath A, Mohanty S, Mohanty P, Gianni C, Della Rocca D, Sabri A, Kim SG, Natale A, Di Biase L. Long-term outcomes of different ablation strategies for ventricular tachycardia in patients with structural heart disease: systematic review and meta-analysis. Europace. 2018 Jan 1;20(1):104-115. doi: 10.1093/europace/eux109. PMID 28575378
- [Background] Wissner E, Stevenson WG, Kuck KH. Catheter ablation of ventricular tachycardia in ischaemic and non-ischaemic cardiomyopathy: where are we today? A clinical review. Eur Heart J. 2012 Jun;33(12):1440-50. doi: 10.1093/eurheartj/ehs007. Epub 2012 Mar 11. PMID 22411192
- [Background] Natale A, Raviele A, Al-Ahmad A, Alfieri O, Aliot E, Almendral J, Breithardt G, Brugada J, Calkins H, Callans D, Cappato R, Camm JA, Della Bella P, Guiraudon GM, Haissaguerre M, Hindricks G, Ho SY, Kuck KH, Marchlinski F, Packer DL, Prystowsky EN, Reddy VY, Ruskin JN, Scanavacca M, Shivkumar K, Soejima K, Stevenson WJ, Themistoclakis S, Verma A, Wilber D; Venice Chart members. Venice Chart International Consensus document on ventricular tachycardia/ventricular fibrillation ablation. J Cardiovasc Electrophysiol. 2010 Mar;21(3):339-79. doi: 10.1111/j.1540-8167.2009.01686.x. Epub 2010 Jan 15. No abstract available. PMID 20082650
- [Background] Tanawuttiwat T, Nazarian S, Calkins H. The role of catheter ablation in the management of ventricular tachycardia. Eur Heart J. 2016 Feb 14;37(7):594-609. doi: 10.1093/eurheartj/ehv421. Epub 2015 Aug 31. PMID 26324538
- [Background] Stevenson WG, Khan H, Sager P, Saxon LA, Middlekauff HR, Natterson PD, Wiener I. Identification of reentry circuit sites during catheter mapping and radiofrequency ablation of ventricular tachycardia late after myocardial infarction. Circulation. 1993 Oct;88(4 Pt 1):1647-70. doi: 10.1161/01.cir.88.4.1647. PMID 8403311
- [Background] Fernandez-Armenta J, Penela D, Acosta J, Andreu D, Evertz R, Cabrera M, Korshunov V, Vassanelli F, Martinez M, Guasch E, Arbelo E, Maria Tolosana J, Mont L, Berruezo A. Substrate modification or ventricular tachycardia induction, mapping, and ablation as the first step? A randomized study. Heart Rhythm. 2016 Aug;13(8):1589-95. doi: 10.1016/j.hrthm.2016.05.013. Epub 2016 May 12. PMID 27180621
- [Background] Cano O, Hutchinson M, Lin D, Garcia F, Zado E, Bala R, Riley M, Cooper J, Dixit S, Gerstenfeld E, Callans D, Marchlinski FE. Electroanatomic substrate and ablation outcome for suspected epicardial ventricular tachycardia in left ventricular nonischemic cardiomyopathy. J Am Coll Cardiol. 2009 Aug 25;54(9):799-808. doi: 10.1016/j.jacc.2009.05.032. PMID 19695457
- [Background] Hutchinson MD, Gerstenfeld EP, Desjardins B, Bala R, Riley MP, Garcia FC, Dixit S, Lin D, Tzou WS, Cooper JM, Verdino RJ, Callans DJ, Marchlinski FE. Endocardial unipolar voltage mapping to detect epicardial ventricular tachycardia substrate in patients with nonischemic left ventricular cardiomyopathy. Circ Arrhythm Electrophysiol. 2011 Feb;4(1):49-55. doi: 10.1161/CIRCEP.110.959957. Epub 2010 Dec 3. PMID 21131557
- [Background] Meng L, Tseng CH, Shivkumar K, Ajijola O. Efficacy of Stellate Ganglion Blockade in Managing Electrical Storm: A Systematic Review. JACC Clin Electrophysiol. 2017 Sep;3(9):942-949. doi: 10.1016/j.jacep.2017.06.006. PMID 29270467